CLINICAL TRIAL: NCT01077817
Title: The Risk of Esophageal Cancer in Relation to the Treatment and Prevention of Osteoporosis in Women
Brief Title: Observational Study of Incidence Rates of Esophageal Cancer in Women Taking Medications for the Prevention or Treatment of Osteoporosis (MK-0217A-352)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Collaborators: World Health Information Science Consultants, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 0217A-352; EP02001.029 (Other: Merck); 2010_015 (Other: Merck)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2013-05-01 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Cancer; Squamous Cell Carcinoma; Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell; Adenocarcinoma | interventions — Alendronate; Etidronic Acid; Ibandronic Acid; Risedronic Acid; Raloxifene Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Esophageal Cancer Cases: Participants with any United Kingdom General Practice Research Database (GPRD) Medical code for esophageal cancer (cases). Cases were confirmed and case onset dates determined by electronic algorithm (based on electronic medical record data) or by medical record review.
  Interventions: Drug: Alendronate; Drug: Etidronate; Drug: Ibandronate; Drug: Risedronate; Drug: Raloxifene
- Comparison Sample (Case-Cohort): Participants who were matched to cases by age and membership in the GPRD on the case's onset date, and had not experienced any form of esophageal cancer or Paget's Disease and had not received oral or intravenous steroids or chemotherapy or radiotherapy, as indicated by GPRD codes.
  Interventions: Drug: Alendronate; Drug: Etidronate; Drug: Ibandronate; Drug: Risedronate; Drug: Raloxifene
- Non-treated Comparators: Participants who did not initiate treatment of osteoporosis with a study drug
- Alendronate: Participants initiating treatment for osteoporosis with alendronate
  Interventions: Drug: Alendronate
- Etidronate: Participants initiating treatment for osteoporosis with etidronate
  Interventions: Drug: Etidronate
- Ibandronate: Participants initiating treatment for osteoporosis with ibandronate
  Interventions: Drug: Ibandronate
- Risedronate: Participants initiating treatment for osteoporosis with risedronate
  Interventions: Drug: Risedronate
- Raloxifene: Participants initiating treatment for osteoporosis with raloxifene
  Interventions: Drug: Raloxifene

INTERVENTIONS:
Drug: Alendronate
  Other Names: FOSAMAX®
  Groups: Alendronate; Comparison Sample (Case-Cohort); Esophageal Cancer Cases
Drug: Etidronate
  Other Names: DIDRONEL®
  Groups: Comparison Sample (Case-Cohort); Esophageal Cancer Cases; Etidronate
Drug: Ibandronate
  Other Names: BONIVA®
  Groups: Comparison Sample (Case-Cohort); Esophageal Cancer Cases; Ibandronate
Drug: Risedronate
  Other Names: ACTONEL®; ATELVIA®
  Groups: Comparison Sample (Case-Cohort); Esophageal Cancer Cases; Risedronate
Drug: Raloxifene
  Other Names: EVISTA®
  Groups: Comparison Sample (Case-Cohort); Esophageal Cancer Cases; Raloxifene

SUMMARY:
This is a 2-phase retrospective database study, using both case-cohort and inception (intention-to-treat) cohort analyses to evaluate any association between oral treatments for osteoporosis and the risk of esophageal cancer in women.

ELIGIBILITY:
Inclusion Criteria:

* Cases:

  * Women in the database aged 55 or older between 1996 and 2008 with diagnosis of esophageal cancer
* Comparator Controls:

  * Each case was matched to all women in the random subcohort of 25,000 who had the same year of birth as the case and were in the database at the time of diagnosis.

Exclusion Criteria:

* Women with diagnosis of any other cancer or Paget's Disease or who have received oral or intravenous steroids before the index date

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have at least two years of experience in the GPRD and are 55 or older between 1996 and 2008; all cases of esophageal cancer were identified and matched to all women in the comparison sample (all women with same year of birth drawn from the random subsample of 25,000).
Sampling Method: Probability Sample
Enrollment: 684815 (Actual)
Dates: Start 2010-02-26 (Actual); Primary Completion 2012-02-16 (Actual); Study Completion 2012-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alec Walker, MD, DrPH, Study Director — World Health Information Science Consultants, LLC

REFERENCES:
- See also: EUPAS Register (EUPAS17909) — http://www.encepp.eu/encepp/viewResource.htm?id=19310

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were not recruited nor enrolled in this study. This study is a retrospective observational study. Data from the GPRD were anonymized and used to develop participant cohorts. All diagnoses and treatments were recorded in the course of routine medical practice.
Pre-assignment Details: 684,815 women in the General Practice Research Database (GPRD) formed the Overall Study Population. These women met the demographic criteria of being age 55 or older, were born between 1922 and 1955, had more than 720 days experience in the GPRD and at least one of those days fell between 1996 and 2008.
Period: Overall Study
Arm/Group | Overall Study Population
Started | 684815 (STARTED and COMPLETED is the number of participants meeting incl./excl. criteria in the GPRD.)
Completed | 684815
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study Population
Number analyzed (Participants) | 684815
Age, Customized [Number; unit: Participants]
  <55 | 0
  ≥55 | 684815
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 684815
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Exposure to Study Drugs (Case-Cohort Analysis)
Description: To determine the use of study drugs (alendronate, etidronate, ibandronate, risedronate, and raloxifene) among female participants with esophageal cancer (cases) and a comparison subcohort, a case-cohort analysis was performed using women meeting criteria from the General Practice Research Database (GPRD, United Kingdom). Exposure to osteoporosis drugs administered 720 days before cancer onset was determined in cases and compared to contemporaneous assessments in a comparison subcohort matched by year of birth and membership in the GPRD on the case's onset date. Cases were confirmed and case onset dates determined by electronic algorithm (based on electronic medical record data) or by medical record review.
Time Frame: Exposure to study drug at least 720 days before disease onset
Population: Case-Cohort analysis population came from the Overall Study Population and comprised 929 women with esophageal cancer (cases) and a Comparison Sample of 338,911 matched control women. Participants may have been exposed to more than one study drug. Also, one comparator may have been used for multiple study drugs.
Measure: Number; unit: Percentage of participants
Groups:
- Esophageal Cancer Cohort: Participants with any GPRD Medical Code for esophageal cancer (cases).
- Comparison Sample (Case Cohort): Participants who were matched to cases by age and membership in the GPRD on the case's onset date, and had not experienced any form of esophageal cancer or Paget's Disease and had not received oral or intravenous steroids or chemotherapy or radiotherapy, as indicated by GPRD codes.
Arm/Group | Esophageal Cancer Cohort | Comparison Sample (Case Cohort)
Number analyzed (Participants) | 929 | 338911
Percentage of participants
  Alendronate | 4.6 | 2.7
  Etidronate | 3.7 | 2.1
  Ibandronate | 0.3 | 0.03
  Risedronate | 2.6 | 0.9
  Raloxifene | 0.3 | 0.4
Statistical Analysis 1: Comparison: Esophageal Cancer Cohort vs Comparison Sample (Case Cohort); A hazard ratio estimate was calculated from the case-control matched set to measure the risk association between exposure to alendronate treatment and incidence of esophageal cancer; Test type: Superiority or Other; Logistic Regression Model; The case-cohort hazard ratio estimate for drug exposure was based on analysis of all cases of esophageal cancer and their comparison sample; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.7 to 1.5]
Statistical Analysis 2: Comparison: Esophageal Cancer Cohort vs Comparison Sample (Case Cohort); A hazard ratio estimate was calculated from the case-control matched set to measure the risk association between exposure to etidronate treatment and incidence of esophageal cancer; Test type: Superiority or Other; Logistic Regression Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.9 to 2.0]
Statistical Analysis 3: Comparison: Esophageal Cancer Cohort vs Comparison Sample (Case Cohort); A hazard ratio estimate was calculated from the case-control matched set to measure the risk association between exposure to ibandronate treatment and incidence of esophageal cancer; Test type: Superiority or Other; Logistic Regression Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 4.9, 95% CI 2-sided [1.4 to 16.7]
Statistical Analysis 4: Comparison: Esophageal Cancer Cohort vs Comparison Sample (Case Cohort); A hazard ratio estimate was calculated from the case-control matched set to measure the risk association between exposure to risedronate treatment and incidence of esophageal cancer; Test type: Superiority or Other; Logistic Regression Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.6, 95% CI 2-sided [1.0 to 2.5]
Statistical Analysis 5: Comparison: Esophageal Cancer Cohort vs Comparison Sample (Case Cohort); A hazard ratio estimate was calculated from the case-control matched set to measure the risk association between exposure to raloxifene treatment and incidence of esophageal cancer; Test type: Superiority or Other; Logistic Regression Model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.2 to 2.2]

2. Primary Outcome: Number of Cases of Esophageal Cancer Per 100,000 Woman-Years (Intent-to-Treat Analysis)
Description: To assess the relative risk of esophageal cancer associated with osteoporosis study drugs (alendronate, etidronate, ibandronate, risedronate, and raloxifene), initiators of osteoporosis drugs and non-initiators (comparators, women sharing match criteria with the initiator) entered an inception cohort for every three-month period, beginning in the first quarter of 1996. Assignment to study drug exposure group remained fixed from the start of follow-up, analogous to an intent-to-treat analysis. The risk of esophageal cancer among initiators of study drug compared to non-initiators of study drug was estimated through calculation of a hazard ratio. For calculation of 721+ day hazard ratios, only esophageal cancer cases occurring at least 721 days from initiation of study drug were used. For calculation of 1441+ day hazard ratios, only esophageal cancer cases occurring at least 1441 days from initiation of study drug were used.
Time Frame: Up to approximately 7.3 years of follow-up
Population: Inception Cohort came from the Overall Study Population beginning treatment with an osteoporosis study drug (initiators, 78,630 women) and 300,610 matched control women, who did not receive study drug (noninitiators). Participants may have been exposed to more than one study drug. Also, one comparator may have been used for multiple study drugs.
Measure: Number; unit: Number of cases per 100,0000 woman-years
Groups:
- Comparators: Participants who did not initiate osteoporosis treatment with a study drug
- Alendronate: Participants who initiated osteoporosis treatment with alendronate
- Etidronate: Participants who initiated osteoporosis treatment with etidronate
- Ibandronate: Participants who initiated osteoporosis treatment with ibandronate
- Risendronate: Participants who initiated osteoporosis treatment with risedronate
- Raloxifene: Participants who initiated osteoporosis treatment with raloxifene
Arm/Group | Comparators | Alendronate | Etidronate | Ibandronate | Risendronate | Raloxifene
Number analyzed (Participants) | 300610 | 48377 | 7851 | 3941 | 15655 | 2806
Number of cases per 100,0000 woman-years | 32 [0.5 to 1.6] | 32 [0.6 to 2.0] | 42 [NA to NA] | 46 [0.4 to 2.5] | 47 [0.2 to 3.9] | 29
Statistical Analysis 1: Comparison: Comparators vs Alendronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of alendronate compared to non-initiators of alendronate. For calculation of this hazard ratio, esophageal cancer cases occurring during the entire follow-up period were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.7 to 1.3]
Statistical Analysis 2: Comparison: Comparators vs Etidronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of etidronate compared to non-initiators of etidronate. For calculation of this hazard ratio, esophageal cancer cases occurring during the entire follow-up period were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.8 to 2.0]
Statistical Analysis 3: Comparison: Comparators vs Ibandronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of ibandronate compared to non-initiators of ibandronate. For calculation of this hazard ratio, esophageal cancer cases occurring during the entire follow-up period were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.5 to 3.4]
Statistical Analysis 4: Comparison: Comparators vs Risendronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of risendronate compared to non-initiators of risendronate. For calculation of this hazard ratio, esophageal cancer cases occurring during the entire follow-up period were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 1.3, 95% CI 2-sided [0.9 to 2.0]
Statistical Analysis 5: Comparison: Comparators vs Raloxifene; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of raloxifene compared to non-initiators of raloxifene. For calculation of this hazard ratio, esophageal cancer cases occurring during the entire follow-up period were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.3 to 2.3]
Statistical Analysis 6: Comparison: Comparators vs Alendronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of alendronate compared to non-initiators of alendronate. For calculation of 721+ day hazard ratios, only esophageal cancer cases occurring at least 721 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.7 to 1.5]
Statistical Analysis 7: Comparison: Comparators vs Etidronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of etidronate compared to non-initiators of etidronate. For calculation of 721+ day hazard ratios, only esophageal cancer cases occurring at least 721 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.7 to 1.9]
Statistical Analysis 8: Comparison: Comparators vs Ibandronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of ibandronate compared to non-initiators of ibandronate. For calculation of 721+ day hazard ratios, only esophageal cancer cases occurring at least 721 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Hazard Ratio (HR) = 3.0, 95% CI 2-sided [0.8 to 11.1]
Statistical Analysis 9: Comparison: Comparators vs Risendronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of risedronate compared to non-initiators of risedronate. For calculation of 721+ day hazard ratios, only esophageal cancer cases occurring at least 721 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Hazard Ratio (HR) = 1.8, 95% CI 2-sided [1.1 to 3.0]
Statistical Analysis 10: Comparison: Comparators vs Raloxifene; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of raloxifene compared to non-initiators of raloxifene. For calculation of 721+ day hazard ratios, only esophageal cancer cases occurring at least 721 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.1 to 2.7]
Statistical Analysis 11: Comparison: Comparators vs Alendronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of alendronate compared to non-initiators of alendronate. For calculation of 1441+ day hazard ratios, only esophageal cancer cases occurring at least 1441 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional Hazards Regression Model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.5 to 1.6]
Statistical Analysis 12: Comparison: Comparators vs Etidronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of etidronate compared to non-initiators of etidronate. For calculation of 1441+ day hazard ratios, only esophageal cancer cases occurring at least 1441 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional hazards regression model — Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.6 to 2.0]
Statistical Analysis 13: Comparison: Comparators vs Risendronate; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of risedronate compared to non-initiators of risedronate. For calculation of 1441+ day hazard ratios, only esophageal cancer cases occurring at least 1441 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional hazards regression model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.4 to 2.5]
Statistical Analysis 14: Comparison: Comparators vs Raloxifene; A hazard ratio was calculated to estimate the risk of esophageal cancer among initiators of raloxifene compared to non-initiators of raloxifene. For calculation of 1441+ day hazard ratios, only esophageal cancer cases occurring at least 1441 days from initiation of study drug (data not shown) were used; Test type: Superiority or Other; Proportional hazards regression model; Year of birth, calendar quarter of cohort entry, and exposure history were stratified in this model; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.2 to 3.9]

ADVERSE EVENTS:
Description: Adverse events were not collected during this study.
Arm/Group | Overall Study Population
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No